CLINICAL TRIAL: NCT05030675
Title: Phase I Open-Label Study of Fostamatinib, a SYK Inhibitor, in Patients With Lower-Risk Myelodysplastic Syndromes or Chronic Myelomonocytic Leukemia Who Have Failed Therapy With Hypomethylating Agents
Brief Title: Fostamatinib for the Treatment of Lower-risk Myelodysplastic Syndromes or Chronic Myelomonocytic Leukemia Who Have Failed Therapy With Hypomethylating Agents
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-1117; NCI-2021-08494 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-1117 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-08-09; First posted 2021-09-01 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Refractory Chronic Myelomonocytic Leukemia; Refractory Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes | interventions — fostamatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (fostamatinib) (Experimental): Patients receive fostamatinib PO BID on days 1-28. Treatment repeats every 28 days for up to 6 cycles (week 24) in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Fostamatinib

INTERVENTIONS:
Drug: Fostamatinib — Given PO
  Other Names: R-935788 Free Acid; R788 Free Acid

SUMMARY:
This phase I trial is to find out the best dose, possible benefits and/or side effects of fostamatinib in treating patients with lower-risk myelodysplastic syndromes or chronic myelomonocytic leukemia who have failed therapy with hypomethylating agents. Fostamatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the safety and tolerability of different doses of fostamatinib in patients with myelodysplastic syndrome (MDS) and chronic myelomonocytic leukemia (CMML) as the measure of adverse events (AEs), serious AEs (SAEs), and laboratory abnormalities on fostamatinib treatment and frequency of discontinuation or interruptions of fostamatinib due to fostamatinib related AEs.

SECONDARY OBJECTIVES:

I. To assess overall survival (OS), duration of response, relapse-free survival (RFS).

II. To assess overall response (OR) rate to different dose schedules of fostamatinib in patients with MDS and CMML following International Working Group (IWG) 2006 response criteria.

III. Hematological response at the end of 2 cycles for each dose level. IV. Frequency of dose escalation of fostamatinib to a dose greater than 100 mg twice daily (BID).

V. Frequency of platelet transfusion independence. VI. Frequency of red blood cell (RBC) transfusion independence for > 8 weeks. VII. Endpoints related to correlative studies.

OUTLINE: This is a dose-escalation study.

Patients receive fostamatinib orally (PO) BID on days 1-28. Treatment repeats every 28 days for up to 6 cycles (week 24) in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years as MDS is a very rare disease in the pediatric setting
* Diagnosis of MDS or CMML according to World Health Organization (WHO) and very low, low or intermediate risk by Revised International Prognostic Scoring System (IPSS-R) (with IPSS-R score of =< 3.5)
* Patients need to have not responded to prior therapy with hypomethylating agents (HMAs). These could include azacitidine, decitabine, SGI-110, ASTX727. Patients will need to have received at least 4 cycles of HMA. Patients with relapse or progression after any number of cycles of HMA by IWG 2006 criteria will also be candidates. Patients with MDS with isolated del(5q) must have received prior therapy with lenalidomide
* Cytopenias, in the form of anemia and thrombocytopenia, as follows:

  * Hemoglobin < 10 g/dL OR
  * Platelets < 75 x10^9/L OR
  * Transfusion dependency, defined as the receipt of any red blood cell or platelet transfusions within at least 28 days prior to the start of study treatment
* Patient (or patient's legally authorized representative) must have signed an informed consent document indicating that the patient understands the purpose of and procedures required for the study and is willing to participate in the study
* Total bilirubin < 2 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 1.5 x ULN
* Serum creatinine clearance > 30 mL/min and no end/stage renal disease (using Cockcroft-Gault)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Hydroxyurea for control of leukocytosis is allowed at any time prior to or during study if considered to be in the best interest of the patient
* Both females of childbearing potential and males with female partners of childbearing potential must agree to use contraception during the study period and for at least one month after the last dose

Exclusion Criteria:

* No prior therapy for MDS or CMML
* Uncontrolled infection not adequately responding to appropriate antibiotics
* Absolute neutrophil count (ANC) < 0.5 x 10^9 k/uL
* Uncontrolled or poorly controlled hypertension, defined as systolic blood pressure >= 135 mmHg or diastolic blood pressure >= 85 mmHg, whether or not the subject is receiving anti-hypertensive treatment
* Female patients who are pregnant or lactating
* Patients with reproductive potential who are unwilling to following contraception requirements (including condom use for males with sexual partners, and for females: prescription oral contraceptives [birth control pills], contraceptive injections, intrauterine devices [IUD], double-barrier method [spermicidal jelly or foam with condoms or diaphragm], contraceptive patch, or surgical sterilization) throughout the study. Reproductive potential is defined as no previous surgical sterilization or females that are not post-menopausal for 12 months
* Female patients with reproductive potential who do not have a negative urine or blood beta-human chorionic gonadotropin (beta human chorionic gonadotropin [HCG]) pregnancy test at screening
* History of an active malignancy within the past 2 years prior to study entry, with the exception of: a. Adequately treated in situ carcinoma of the cervix uteri b. Adequately treated basal cell carcinoma or localized squamous cell carcinoma of the skin or any other malignancy with a life expectancy of more than 2 years
* Patients receiving any other concurrent investigational agent or chemotherapy, radiotherapy, or immunotherapy (within 14 days of initiating study treatment)
* Evidence of graft versus host disease or prior allo-stem cell transplantation within 6 months of Cycle 1 Day 1 or receiving immunosuppressants following a stem-cell procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-08-13 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2024-08-08 (Actual)

PRIMARY OUTCOMES:
The PI doesnt wish to add any Outcome Measures this will be add at the time of results | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo M Bravo, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States